CLINICAL TRIAL: NCT05619003
Title: A Prospective Single-arm Study Investigating the Safety of Biatain Silicone Sacral While Used as Prevention in Hospital-admitted Patients at Risk of Developing a Pressure Injury
Brief Title: Biatain Silicone Sacral for Pressure Injury Prevention in Hospital-admitted Patients at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP346
Record Dates: First submitted 2022-11-04; First posted 2022-11-16 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pressure Injury Prevention

STUDY DESIGN:
Intervention Model Description: Open-labelled, non-comparative, single-arm, prospective, multi-center investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biatain Silicone Sacral Dressing (Experimental)
  Interventions: Device: Biatain Silicone Sacral dressing

INTERVENTIONS:
Device: Biatain Silicone Sacral dressing — Biatain Silicone Sacral dressing will be applied over the bony prominence of the sacral area as part of a PIP (Pressure Injury Prevention) protocol in patients at risk

SUMMARY:
A post market clinical follow-up study investigating the safety of Biatain Silicone Sacral while used as prevention in hospital admitted patients at risk of developing a pressure injury.

DETAILED DESCRIPTION:
The investigation was a multi-centre, open label, non-comparative, single-arm, prospective study, conducted at three investigational sites in Danish hospitals. 67 hospital-admitted patients were enrolled in the study over a 3-month recruitment period. The target population were patients ≥18 years of age with an expected hospital-stay of more than 24 hours from baseline and a Braden score of 6-18.

At daily visits skin inspections for signs of non-blanchable erythema or sacral pressure injury were performed by partial lift and reapplication of the dressing. After 7 days, or earlier if the patient was discharged, a termination visit was performed. Skin assessment was performed upon removal of the dressing and a termination form completed. Information regarding adverse events and device deficiencies were collected at all visits.

There were no follow-up visits after termination of the study.

ELIGIBILITY:
Inclusion Criteria:

* Hospital-admitted patients at risk of developing a pressure injury with an expected hospital-stay of more than 24 hours from visit 1
* ≥18 years of age and has full legal capacity
* Has given written consent to participate by signing the Informed Consent signature Form
* Has a Braden score of 6-18 at screening (performed within the last 24 hours)
* Intact sacral skin (non-breached skin, without signs of non-blanchable erythema over bony prominence/pre-existing sacral pressure injury over bony prominence)

Exclusion Criteria:

* Suspected or actual spinal injury precluding the patient from being turned
* Sacral erythema, sacral pressure marks, pre-existing sacral pressure injury
* Trauma to sacrum
* Topical treatment with steroid creme in the sacral area (treatment must have been terminated at least 14 days prior to enrollment)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Overgaard, SSM, Study Chair — Coloplast A/S
Locations (3):
- Denmark (3):
  - Bispebjerg Hospital, Copenhagen
  - Herlev Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Biatain Silicone Sacral Dressing: Biatain Silicone Sacral will be applied over the bony prominence of the sacral area
Period: Overall Study
Arm/Group | Biatain Silicone Sacral Dressing
Started | 67
Completed | 66
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Numbers of participants constitutes the ITT population (participants exposed to the investigational device with information on at least one endpoint) and differ from the overall (safety population constituted by all subjects with a valid informed consent)
Arm/Group | Biatain Silicone Sacral Dressing
Number analyzed (Participants) | 66
Age, Continuous [Mean (Full Range); unit: years] | 70.5 [46 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 66
BMI [Mean (Full Range); unit: kg/m2] | 27.4 [15 to 50]
Urinary incontinence [Count of Participants; unit: Participants] | 18
Faecal incontinence [Count of Participants; unit: Participants] | 12
Braden Scale Score [Mean (Full Range); unit: scores on a scale] — The Braden Scale is a standardized assessment tool used in healthcare to assess a patient's risk for developing pressure injuries. The total Braden Scale score ranges from 6 to 23, with lower scores indicating higher susceptibility to pressure ulcers
  scores on a scale | 15.9 [11 to 18]

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Evaluate the safety of Biatain Silicone Sacral. Adverse events considered related to the investigational device by the investigator during the investigation period (up to 7 days or until discharged)
Time Frame: 7 days
Measure: Number; unit: Adverse events
Arm/Group | Biatain Silicone Sacral Dressing
Number analyzed (Participants) | 67
Adverse events | 0

2. Secondary Outcome: Number of Device Deficiencies
Description: Evaluate the safety of Biatain Silicone Sacral. Number of device deficiencies during the investigation period (up to 7 days or until discharged)
Time Frame: 7 days
Measure: Number; unit: Device deficiencies
Groups:
- Biatain Silicone Sacral Dressing: Biatain Silicone Sacral dressing will be applied over the bony prominence of the sacral area
Arm/Group | Biatain Silicone Sacral Dressing
Number analyzed (Participants) | 67
Device deficiencies | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (day 1, visit 1) and at all daily visits until termination visit (latest after 7 days). There was no follow-up after study termination.
Groups:
- Biatain Silicone Sacral Dressing: 67 patients were treated with Biatain Silicone Sacral dressing over the bony prominence of the sacral area as part of a pressure injury prevention protocol
Arm/Group | Biatain Silicone Sacral Dressing
All-Cause Mortality (participants affected / at risk) | 1/67
Serious Adverse Events (participants affected / at risk) | 4/67
Other Adverse Events (participants affected / at risk) | 5/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biatain Silicone Sacral Dressing (N=67)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 — Worsening of shortness of breath. Event assessed as not related to the investigational device by the investigator
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Patient admitted with end stage cirrhosis or cancer of the liver. Event assessed as not related to the investigational device by the investigator
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — Aspiration to the lungs in conjunction with gastroscopy. Event assessed as not related to the investigational device by the investigator
Intraabdominal bleeding (Surgical and medical procedures) | 1 — patient experienced intraabdominal bleeding following a total colectomy due to ulcerative colitis. Event assessed as not related to the investigational device by the investigator
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biatain Silicone Sacral Dressing (N=67)
Incision site pain (Nervous system disorders) | 5 (5) — All events assessed as not related to the investigational device by the investigator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT05619003/Prot_SAP_000.pdf